CLINICAL TRIAL: NCT07371988
Title: Efficacy of Narrative Therapy for Older People With Depression
Acronym: NTOPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HU-STA-00001793; 9231614 (Other: City University of Hong Kong)
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Depression
Keywords: Randomized controlled trial; Depressive Disorders; Narrative Therapy group; Self-stigma; Hope; Wellbeing
MeSH Terms: conditions — Depression; Depressive Disorder | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants in the intervention group will receive an narrative therapy group in addition to treatment as usual provided by the elderly centre such as interest classes and recreational activities. Narrative therapy group consists 8 session, with one session will be conducted per week, with each session lasting for about 90 minutes. A social worker and a counsellor will be recruited to run narrative groups at collaborative elderly centres. The narrative therapy group provides the following intervention strategies: engagement, de-construction, re-construction, and co-construction of personal identities. Standardized program manual of this narrative group will be developed by the research team. The social workers delivering the narrative therapy group in this project will receive the program manuals, training and supervision from the project team and an experienced clinical psychologist to ensure that the intervention groups follow the program manual.
Who Masked: Investigator
Masking Description: A research assistant, who is not involve in the randomized allocation of participants and delivery of intervention group, will conduct pre- and post-intervention outcome assessments using standardised assessment tools.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8-session narrative therapy group (Active Comparator): This study includes a two arms parallel groups for comparison. Participants in the intervention group will receive an eight-session narrative therapy group in addition to treatment as usual provided by the elderly centres such as interest classes and recreational activities. The narrative therapy group will be conducted by an experienced and trained social worker and counselor.
  Interventions: Behavioral: Narrative therapy group
- Waitlist Control (Other): Waitlist control group will receive will receive treatment as usual provided by the elderly centre, including recreational activities and interest classes, at the initial stage and will receive a brief narrative therapy program at a later stage
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Narrative therapy group — Narrative therapy group consists of 8 sessions, with one session will be conducted per week, with each session lasting for about 90 minutes. A social worker and a counsellor will be recruited to run narrative groups at collaborative elderly centres. The narrative therapy group provides the following intervention strategies: engagement, de-construction, re-construction, and co-construction of personal identities. A standardized program manual of this narrative group will be developed by the research team. The social workers delivering the narrative therapy group in this project will receive the program manuals, training and supervision from the project team and an experienced clinical psychologist to ensure that the intervention groups follow the program manual.
  Arms: 8-session narrative therapy group
Other: Treatment as usual (TAU) — Waitlist control group will receive will receive treatment as usual provided by the elderly centre, including recreational activities and interest classes, at the initial stage and will receive a brief narrative therapy program at a later stage
  Arms: Waitlist Control

SUMMARY:
The research aims to investigate the efficacy of a narrative therapy group in reducing depressive symptoms among older people.

This study adopts a mixed methods research design, involving both quantitative and qualitative approaches. In the quantitative study, a randomised controlled trial will compare a narrative therapy group with a waitlist control group to determine whether an eight-session narrative therapy group can reduce depressive symptoms in older people. The eight-session narrative therapy group will be delivered by a trained and experienced social worker or counsellor, and intervention outcomes will be assessed before and after the intervention using a standardised assessment tool for depressive symptoms. The qualitative study aims to examine the benefits, advantages, and limitations of the narrative therapy group from the users' perspective.

DETAILED DESCRIPTION:
Efficacy of Narrative Therapy for older people with depression

Objective: This research aims to investigate the efficacy of a narrative therapy group in reducing depressive symptoms among older people.

Research Method: This study adopts a mixed methods research design, involving both quantitative and qualitative approaches. Using a randomised controlled trial, the quantitative study aims to investigate the effectiveness of a narrative therapy group in reducing self-stigma among people with depression. The qualitative study aims to examine the benefits, advantages, and limitations of the narrative therapy group from the users' perspective. Ethical considerations were reviewed and approved by the Research Committee of the City University of Hong Kong [Reference No.: HU-STA-00001793]. Written informed consent will be obtained from each participant on the day of initial screening for eligibility.

Quantitative Research Method

Objective. This quantitative study aims to investigate the effectiveness of the narrative therapy group in reducing depressive symptoms among older people.

Research Design. This study is a multicentre randomised waitlist control trial. Eligible participants will be recruited from local elderly centres in various districts, through open recruitment via promotional activities and referrals from these centres. Recruitment will take place over the study period. Using block randomisation, participants will be randomly assigned in a 1:1 ratio to either the intervention group or the waitlist control group. Participants in the intervention group will receive an eight-session narrative therapy group in addition to treatment as usual, while those in the waitlist control group will receive treatment as usual provided by the elderly centre. A research assistant, blinded to group allocation, will conduct pre- and post-intervention outcome assessments using standardised assessment tools.

Hypotheses: After completing the narrative therapy group, participants will show significantly greater improvement in depressive symptoms, self-esteem, self-stigma, sense of hope and wellbeing at post-intervention.

Subject inclusion and exclusion criteria. The inclusion criteria are:

1. aged 60 years or above;
2. exhibiting depressive symptoms as assessed using a standardised assessment tool, namely the Chinese Beck Depression Inventory-II (BDI; Byrne et al., 2004), with a BDI score between 10 and 30;
3. being a service user of an elderly centre; and
4. providing informed consent to participate in this research.

Exclusion criteria

1. Individuals with severe depression (i.e. a BDI score ≥ 31), dementia, psychosis, or self-reported suicidal thoughts are excluded from this study.
2. Individuals currently receiving a therapeutic intervention are also not excluded from this study.

Sample Size Estimation. The sample size of this study is estimated by using power analysis G*Power 3.1. Studies on interventions report a small to medium effect size in reducing depressive symptoms. This study aims to detect a medium effect size (i.e., Cohen's d = 0.5) with a statistical power of 0.80 for all intervention outcomes. A minimum sample size of 82 participants is required. Considering a dropout rate of 25%, a total of 110 participants will be recruited.

Intervention group. Narrative therapy group consists 8 session, with one session will be conducted per week, with each session lasting for about 90 minutes. A social worker and a counsellor will be recruited to run narrative groups at collaborative elderly centres. A standardized program manual is designed by the research team. The narrative therapy group provides the following intervention strategies: engagement, de-construction, re-construction, and co-construction of personal identities. In the deconstruction phase (sessions 2-3), externalising conversation is used to separate the person from the problem. In the reconstruction of an alternative new identity (sessions 4-5), unique life experiences that do not fit self-stigmatising beliefs are identified, facilitating the development of a new perspective on one's life story. In addition, the technique of re-membering is used to help participants reconnect with trustworthy individuals, such as teachers, relatives, and peers, who can provide alternative perspectives and recognition of participants' strengths, values, character, and resources. Finally, in the co-construction of new alternative self-identities (sessions 6-8), a definitional ceremony is conducted to invite others, such as family members, to recognise and affirm the person's new positive self-identity.

Waitlist control group. The waitlist control group will receive treatment as usual provided by the elderly centre, including recreational activities and interest classes, at the initial stage and will receive a brief narrative therapy program at a later stage.

Outcome assessment tools. The primary outcome is the reduction of depressive symptoms, assessed by the Chinese Beck Depression Inventory-II (BDI). BDI is a 21-item scale to assess self-reported depression. The severity scale is as follows: a score of 0-13 represents minimal or no depression; 14-19 indicates mild depression; 20-28 indicates moderate depression; and 29-63 indicates severe depression. A cut-off point of a BDI score ≥ 14 was adopted in this study as indicative of clinical depression.

Secondary outcomes include improvements in self-stigma, self-esteem, hope and wellbeing, which are assessed by the following standardized scales.

The Chinese Internalised Stigma of Mental Illness (ISMI; Young et al., 2017) is a 10 -item self-reported scale to measure changes in self-stigma.

The Chinese Rosenberg Self-Esteem Scale (RSES; Peng et al., 2024) is a 10-item scale to assess participants' self-reported self-esteem.

The Chinese Dispositional Hope Scale (DHS; Sun et al., 2012) is a 12-item scale used to assess participants' self-reported hope.

The Chinese WHO 5-item Well-Being Index (WHO-5; Fung et al., 2022) is a 5-item scale for assessing subjective wellbeing.

Data analysis. An analysis will be performed in accordance with the intent-to-treat principle using multiple imputation for any missing data. For all analyses, two-tailed p values of < 0.05 is considered statistically significant. Data analyses will be performed using SPSS 29.0. Within group intervention effects are investigated using paired-sample t-tests. Between group intervention effects are investigated using a 2 (group) x 2 (time) repeated measures one-way analysis of variance (ANOVA). Within and between group effect sizes are computed using Cohen's d, with values of 0.2, 0.5, and 0.8 considered small, medium, and large respectively (Cohen, 1988).

Fidelity of intervention. Standardized program manual of this narrative group will be developed by the research team. The social workers delivering the narrative therapy group in this project will receive the program manuals, training and supervision from the project team and an experienced clinical psychologist to ensure that the intervention groups follow the program manual.

Qualitative Research Method

Objective. This qualitative study aims to explore the benefits, advantages and limitations of the narrative therapy group from the users' perspective.

Research Design. The qualitative study uses an interpretative interview method with purposive sampling. In-depth interviews and focus group will be conducted with 15 intervention group participants, with each interview lasting approximately 90 minutes.

Data collection. Each in-depth interview and focus group will be facilitated by a research staff with an interview protocol developed for this study. Participants will be asked questions such as: "In what ways, if any, did the intervention group help you to reduce your self-stigma?"; "In what ways, if any, did the intervention group help you to improve your mental health such as depression and anxiety"; "In what ways, if any, did the intervention group help you to improve your wellbeing such as improving self-esteem, reducing self-stigma, and building up a sense of hope?"; "What are the advantages and limitations, if any, of the intervention group?"; "and "Any suggestions, if any, for improving the intervention group?". The results of the qualitative analysis will provide insights for further development and modification of the narrative therapy group.

Data analysis. The content of the in-depth interviews and focus groups will be audio-recorded and transcribed into verbatim by the research team. All transcripts of the focus groups will be imported and coded for data management and analysis. Reflective thematic analysis will be used to identify, analyse and report themes so that themes can be developed both inductively (i.e. data-driven) and deductively (i.e. theory-driven). The research team will systematically read and re-read the transcripts, following the six stages of analysis, including: (1) becoming familiar with the data, (2) generating codes, (3) constructing themes, (4) reviewing potential themes, (5) defining and naming themes, and (6) producing the report. Two research staff compare, review and refine the codes, categories and themes until they reach agreement.

ELIGIBILITY:
Inclusion Criteria:

1. aged 60 years or above;
2. exhibiting depressive symptoms as assessed using a standardised assessment tool, namely the Chinese Beck Depression Inventory-II (BDI; Byrne et al., 2004), with a BDI score between 10 and 30;
3. being a service user of an elderly centre; and
4. providing informed consent to participate in this research.

Exclusion Criteria:

1. Individuals with severe depression (i.e. a BDI score ≥ 31), dementia, psychosis, or self-reported suicidal thoughts are excluded from this study; and
2. Individuals currently receiving a therapeutic intervention are not excluded from this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Chinese Beck Depression Inventory-II (BDI) | Before and after the 8-week intervention
  BDI is a 21-item scale with excellent validity, and reliability (Cronbach's α = 0.91), used to assess self-reported depression. The severity scale is as follows: a score of 0-13 represents minimal or no depression; 14-19 indicates mild depression; 20-28 indicates moderate depression; and 29-63 indicates severe depression. A cut-off point of a BDI score ≥ 14 was adopted in this study as indicative of clinical depression. Each item (e.g. Past failure) is rated on a 4-point scale with scores ranging from "0" to "3". The scores are summed over the items, with higher scores indicating a higher severity of symptoms

SECONDARY OUTCOMES:
Chinese Internalised Stigma of Mental Illness (ISMI) | Before and after the 8-weeks intervention.
  The Chinese Internalised Stigma of Mental Illness (ISMI; Young et al., 2017b) is a 10 -item self-reported scale to measure changes in self-stigma in four dimensions, i.e. shame/alienation (ISMI-SH), stereotype endorsement (ISMI-SE), perceived discrimination (ISMI-PD) and social withdrawal (ISMI-SW), with good validity and reliability (Cronbach's α = 0.93; 0.85; 0.75; 0.84 and for ISMI total scale, ISMI-SH, ISMI-SE, ISMI-PD, ISMI-SW). Each item (e.g. People discriminate against me because I have a mental illness) is rated on a 4-point scale from "1" (strongly agree) to "4" (strongly disagree). Scores are averaged over the items, with higher scores indicating greater self-stigma.
Chinese Rosenberg Self-Esteem Scale (RSES) | Before and after the 8-weeks intervention
  The Chinese Rosenberg Self-Esteem Scale (RSES; Leung & Wong, 2008) is a 10-item scale to assess participants' self-reported self-esteem in two dimensions, i.e. self-worth (RSES-SW) and self-depreciation (RSES-SD) with good validity and reliability (Cronbach's α = 0.63; 0.74, and 0.81 for RSES, RESE-SW, and RSES-SD). Each item (e.g. I feel that I have a number of good qualities) is rated on a 4-point scale from "1" (strongly agree) to "4" (strongly disagree). Scores are summed over the items, with higher scores indicating better self-esteem
The Chinese Dispositional Hope Scale (DHS) | Before and after the 8-weeks intervention
  The Chinese Dispositional Hope Scale (DHS; Sun et al., 2012) is a 12-item scale used to assess participants' self-reported hope in tow dimensions, i.e., agency (i.e., goal-directed energy) and pathways (i.e., planning to accomplish goals) with good validity and reliability (Cronbach's α = 0.81; 0.70 and 0.76 for the Hope total scale, agency subscale and pathway subscale). Each item (e.g. I can think of many ways to get out of a jam) is answered using a 4-point scale ranging from "1" (definitely false) to "4" (definitely true). Scores are summed over the items, with higher scores indicating a higher level of hope.
The Chinese WHO 5-item Well-Being Index (WHO-5) | Before and after the 8-weeks intervention
  The Chinese WHO 5-item Well-Being Index (WHO-5; Fung et al., 2022) is a 5-item scale for assessing subjective wellbeing with satisfactory validity and internal consistency (Cronbach's α = 0.85; Fung et al., 2022). Each item (e.g., feel a sense of companionship in life) is rated on a 5-point Likert-type scale ranging from 1 (very dissatisfied) to 5 (very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Kim-wan Daniel Young, PhD, Principal Investigator — City University of Hong Kong
Locations (1):
- City University of Hong Kong, Kowloon Tong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cohen, J. (1988). Statistical power analysis for the behavioral sciences (2nd ed.). Lawrence Erlbaum Associates
- [Background] Lee SW, Stewart SM, Byrne BM, Wong JP, Ho SY, Lee PW, Lam TH. Factor structure of the Center for Epidemiological Studies Depression Scale in Hong Kong adolescents. J Pers Assess. 2008 Mar;90(2):175-84. doi: 10.1080/00223890701845385. PMID 18444112
- [Background] Madigan, S. (2019). Narrative Therapy (2nd edition). American Psychological Association
- [Background] White, M. (2007). Maps of Narrative Practice. W. W. Norton & Company
- [Background] Young, D. K. W., Ng, P. Y., Pan, J. Y., & Cheng, D. (2017b). Validity and reliability of internalized stigma of mental illness (Cantonese). Research on Social Work Practice, 27(1), 103-110. https://doi.org/10.1177/1049731515576209
- [Background] Sun, Q., Ng, K.-M., & Wang, C. (2012). A validation study on a new Chinese version of the Dispositional Hope Scale. Measurement and Evaluation in Counseling and Development, 45(2), 133-148. https://doi.org/10.1177/0748175611429011
- [Background] Peng W, Zhou Y, Chu J, Liu Z, Zheng K, Yao S, Yi J. Factorial and Criterion Validities of the Chinese Version of Rosenberg Self-Esteem Scale Among Undergraduate Students. Psychol Res Behav Manag. 2024 Dec 5;17:4135-4144. doi: 10.2147/PRBM.S494452. eCollection 2024. PMID 39654814
- [Background] Lamarca M, Espinosa V, Acuna V, Vila-Badia R, Balsells-Mejia S, Moritz S, Berna F, Konig C, Gaweda L, Group P, Barajas A, Ochoa S. Reducing self-stigma in psychosis: A systematic review and meta-analysis of psychological interventions. Psychiatry Res. 2024 Dec;342:116262. doi: 10.1016/j.psychres.2024.116262. Epub 2024 Nov 16. PMID 39549598
- [Background] Fung SF, Kong CYW, Liu YM, Huang Q, Xiong Z, Jiang Z, Zhu F, Chen Z, Sun K, Zhao H, Yu P. Validity and Psychometric Evaluation of the Chinese Version of the 5-Item WHO Well-Being Index. Front Public Health. 2022 Mar 30;10:872436. doi: 10.3389/fpubh.2022.872436. eCollection 2022. PMID 35433612